CLINICAL TRIAL: NCT07195552
Title: Clinical Trail: Rapid Immune Modulating Effects
Brief Title: Clinical Trial: Rapid Immune Modulating Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 171-003
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, crossover design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crossover group 1, randomized (Experimental): Crossover study: Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 4 weeks. The order of interventions for this group is A, B, C, D.
  Interventions: Dietary Supplement: Agaricus blazei; Dietary Supplement: Reishi; Dietary Supplement: Turkey Tail; Other: Placebo
- Crossover group 2, randomized (Experimental): Crossover study: Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 4 weeks. The order of interventions for this group is B, D, A, C.
  Interventions: Dietary Supplement: Agaricus blazei; Dietary Supplement: Reishi; Dietary Supplement: Turkey Tail; Other: Placebo
- Crossover group 3, randomized (Experimental): Crossover study: Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 4 weeks. The order of interventions for this group is C, A, D, B.
  Interventions: Dietary Supplement: Agaricus blazei; Dietary Supplement: Reishi; Dietary Supplement: Turkey Tail; Other: Placebo
- Crossover group 4, randomized (Experimental): Crossover study: Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 4 weeks. The order of interventions for this group is D, B, A, C.
  Interventions: Dietary Supplement: Agaricus blazei; Dietary Supplement: Reishi; Dietary Supplement: Turkey Tail; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Agaricus blazei — Agaricus blazei mushroom capsules. 2000 mg per serving
Dietary Supplement: Reishi — Reishi mushroom capsules. 2000 mg per serving.
Dietary Supplement: Turkey Tail — Turkey tail mushroom capsules. 2000 mg per serving.
Other: Placebo — Placebo

SUMMARY:
The goal for this clinical trial is to compare the immune effects of three different medicinal mushrooms to a placebo. The mushrooms include Agaricus, Reishi, and Turkey Tail.

DETAILED DESCRIPTION:
The goal for this clinical trial is to compare acute immune effects of three different medicinal mushrooms to a placebo in a healthy population. The mushrooms include Agaricus, Reishi, and Turkey Tail.

The outcomes include immune cell communication via pro- and anti-inflammatory cytokines, increased immune cell alertness, and immune cell trafficking and surveillance.

These activities happen normally as part of our immune system's circadian cycles and can be significantly enhanced by consuming nutraceutical products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:
* Maintaining a consistent diet and lifestyle routine throughout the study,
* Consistent habit of bland breakfasts on days of clinic visits,
* Abstaining from exercising and nutritional supplements on the morn ing of a study visit,
* Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
* Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Immune Communication | 2 hours after consuming a test product for this study protocol
  Changes to serum cytokine levels. The testing involves a broad panel of pro- and anti-inflammatory cytokines, anti-viral peptides, and regenerative growth factors, using a 27-plex Luminex magnetic bead array and the MagPix® multiplexing system. The following cytokines are tested: IL-1beta, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, eotaxin, basic FGF, G-CSF, GM-CSF, IFN-gamma, IP-10, MCP-1 (MCAF), MIP-1alpha, MIP-1beta, PDGF-BB, RANTES, TNF-alpha, and VEGF.

SECONDARY OUTCOMES:
Immune Cell Surveillance | 2 hours after consuming a test product for this study protocol
  Documentation of changes in immune cell trafficking, i.e., the changes in immune cell numbers in the peripheral blood following administration. Data is collected as 'cell numbers per uL whole blood' for the following immune cell types:
  * Monocytes
  * NK cells
  * NKT cells
  * T cells
  * non-NK nonT cells

OTHER OUTCOMES:
Immune responsiveness | 2 hours after consuming a test product for this study protocol
  Immune cell activation status:
  Observation of immune cell status of alertness, i.e., the changes in the expression of CD25 and CD69. Data is collected as 'mean fluorescence intensity' for the following immune cell types:
  * Monocytes
  * NK cells
  * NKT cells
  * T cells
  * nonNK nonT cells.
  Immune challenges ex vivo:
  Effect on anti-bacterial and anti-viral immune defense activity

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No